CLINICAL TRIAL: NCT00202735
Title: Does Immobilization of the Shoulder in External Rotation Reduce the Recurrence Rate of Shoulder Dislocation?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other); Haukeland University Hospital (Other); Sykehuset i Vestfold HF (Other); Helse Stavanger HF (Other Government); Sykehuset Telemark (Other Government); Sykehuset Buskerud HF (Other); Blefjell Hospital HF (Other Government); Sykehuset Asker og Baerum (Other); St. Olavs Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Svein Svenningsen Dr.med, Sorlandet hospital HF
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 811327
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2005-01

CONDITIONS: Shoulder Dislocation
Keywords: shoulder dislocation; anterior; traumatic; primary; first time; initial; immobilization; external; rotation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immobilization in internal rotation (Active Comparator): Immobilization in internal rotation:All patients in this group are immobilized with the arm in internal rotation.
  The arm is immobilized with a normal collar and cuff device.
  Interventions: Procedure: immobilization in internal rotation
- Immobilization in external rotation. (Experimental): Immobilization in external rotation (ER. All patients in the ER group use a prefabricated shoulder immobilizer (Don Joy Ultrasling ER, 15˚ version.To control the position, a line at the top of the immobilizer is to be parallel with the frontal plane when the arm is correctly placed
  Interventions: Procedure: Arm1:Immobilization in external rotation

INTERVENTIONS:
Procedure: Arm1:Immobilization in external rotation — Immobilization in external rotation (ER) All patients in the ER group use a prefabricated shoulder immobilizer (Don Joy Ultrasling Er,15˚ version).To control the position,a line at the top of the immobilizer is to be parallel with the frontal plane when the arm is correctly placed in 15 degrees of external rotation.
  Other Names: Immobilization in external rotation.
  Arms: Immobilization in external rotation.
Procedure: immobilization in internal rotation — All the patients in the internal rotation(IR) group are immobilized with their arm/shoulder in internal rotation by using a normal collar and cuff device.
  Arms: Immobilization in internal rotation

SUMMARY:
Dislocation of the glenohumeral joint is the most common traumatic joint dislocation. The usual treatment of first time traumatic anterior dislocation of the shoulder is reduction followed by immobilization in a sling for a period of one to three weeks. The incidence of recurrence is high and age at the time of primary dislocation is the chief prognostic factor in determining the risk of recurrence. There is no agreement according to the effect of immobilization,neither to the length of immobilization time. The Bankart lesion with avulsion of the inferior-anterior capsulolabral complex is almost invariably present in patients with anterior shoulder dislocation. Recent and ongoing studies by Eijii Itoi et al,Akita university Japan, gives evidence of the immobilization with the arm held in external rotation may reduce the risk of subsequent instability by approximating the Bankart lesion to the neck of the glenoid giving a more anatomical healing. We have started a prospective randomized study. The patients are assigned to two groups with informed consent. One group are immobilized in internal rotation for 3 weeks and the second group are immobilized in external rotation for 3 weeks. We will compare the rate of relaxation between the groups. Because age is the main prognostic factor we use stratified randomization with two age groups: One group of patients aged between 16 and 24 years and one group aged between 25 and 40 years.The time of observation after initial treatment will be 2 years with follow up after 4 and 10 years. Eleven hospitals and two primary trauma care centers in Norway participate in the study. A subgroup of 50 patients are also planned to be examined with CT and MRI.

DETAILED DESCRIPTION:
See earlier protocol in 2005

ELIGIBILITY:
Inclusion Criteria:

The patient has a first time traumatic anterior dislocation of the shoulder. The dislocation is verified by x-ray examination. The patient is aged between 16 and 40 years.

-

Exclusion Criteria:

An osseous defect of the anterior glenoid rim in which the length is at least 20% and the width at least 1/3 of the the length of the anterior bony glenoid rim.

A fracture of tuberculum majus which do not fall into place after manually reduction of the dislocated shoulder.(That means more than 1 cm diastase)

Damage of the axillary nerve or plexus

The patient is not able to or willing to participate in the study. -

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2005-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reluxation | After 2 years

SECONDARY OUTCOMES:
Function,WOSI score,SIQ score | Between second and third year after the primary dislocation.
Pain,Wosi score and SIQ score | Between the second and third year after the primary dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Svein Svenningsen, M.D., Study Chair — Sorlandet Hospital